CLINICAL TRIAL: NCT04304209
Title: Pd1 Antibody Sintilimab ± Chemoradiotherapy for Locally Advanced Rectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2019-149
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer Stage II; Colorectal Cancer Stage III
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Capecitabine; sintilimab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): After 4 cycles of neoadjuvant sintilimab treatment, the patients and doctors could choose one of the following treatments: (1) surgery, followed by 4 cycles of adjuvant sintilimab with or without Capeox chemotherapy; (2) another 4 cycles of sintilimab, followed by radical surgery or observation (only for patients with clinical complete response).
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Sintilimab; Procedure: total mesorectal excision; Other: Watch and wait
- Cohort B-arm 1 (Experimental): After four cycles of neoadjuvant Sintilimab, Capeox and radiotherapy, the patients and doctors could choose one of the following treatments: (1) curative surgery and four cycles of adjuvant Capeox chemotherapy;(2)four cycles of Capeox chemotherapy then observation (only for patients with clinical complete response after neoadjuvant therapy)
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Sintilimab; Radiation: radiotherapy; Procedure: total mesorectal excision; Other: Watch and wait
- Cohort B-arm 2 (Active Comparator): After four cycles of neoadjuvant Capeox chemotherapy and radiotherapy, the patients and doctors could choose one of the following treatments: (1) curative surgery and four cycles of adjuvant Capeox chemotherapy;(2)four cycles of Capeox chemotherapy then observation (only for patients with clinical complete response after neoadjuvant therapy)
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Radiation: radiotherapy; Procedure: total mesorectal excision; Other: Watch and wait

INTERVENTIONS:
Drug: Oxaliplatin — 130mg/m2, d1 q3w, in Capeox regimen (100mg/m2 when used cocurrently with radiotherapy), intravenous infusion
Drug: Capecitabine — 1000mg/m2, bid, qd1-14, q3w, in Capeox regimen, oral administration
Drug: Sintilimab — 200mg, d1 q3w, intravenous infusion
  Arms: Cohort A; Cohort B-arm 1
Radiation: radiotherapy — neoadjuvant radiotherapy with 50Gy to GTV, 45Gy to CTV in 25 fractions.
  Arms: Cohort B-arm 1; Cohort B-arm 2
Procedure: total mesorectal excision — total mesorectal excision after neoadjuvant treatment
Other: Watch and wait — Watch and wait for cCR patients after neoadjuvant treatment

SUMMARY:
In this study, participants with locally advanced rectal cancer patients will be treated according to MMR/MSI status. There will be two cohorts in this study: Cohort A and Cohort B. For Cohort A, dMMR or MSI-H patients will receive 4 cycles of neoadjuvant Pd1 antibody Sintilimab,followed by one of the following treatments: (1) surgery and adjuvant treatment, (2）another 4 cycles of sintilimab, followed by radical surgery or observation (only for cCR) . For Cohort B, pMMR/MSS/MSI-L patients will be randomized to receive neoadjuvant chemoradiotherapy ± four cycles of Pd1 antibody Sintilimab，followed by one of the following treatments: (1) curative surgery and four cycles of adjuvant chemotherapy;(2)four cycles of chemotherapy then observation (only cCR after neoadjuvant therapy)

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven colorectal adenocarcinoma;
2. Cohort 1: Biopsy tissues with IHC indicates deficient mismatch repair(dMMR),that is,the loss of at least one of the four proteins ,MSH1,MSH2,MSH6,PMS2;or gene detection implies MSI-H; Cohort 2: Biopsy tissues with IHC indicates proficient mismatch repair(pMMR),that is positivity of all four proteins ,MSH1,MSH2,MSH6,PMS2;or gene detection implies MSS/MSI-L
3. Clinical stage for rectal cancer patients is cT3-4N0M0 or cTxN+M0;
4. Preoperative staging methods: all patients need to accept digital rectal examination(DRE).Patients with rectal cancer undergo high-resolution MRI±ultrasound colonoscopy/transrectal ultrasound for preoperative staging. Perienteric lymph nodes with short diameter ≥10mm or the shape of lymph nodes and its MRI characteristics are consistent with typical lymph node metastasis. If endoscopic ultrasonography is used in combination, and there is a contradiction between staging methods, the data should be submitted to the evaluation team of our center for the accurate staging;
5. No symptoms of ileus; or ileus is alleviated after proximal colostomy.
6. No rectal surgery except preventative stoma;
7. No chemotherapy or radiotherapy;
8. No biotherapy (e.g.monoclonal antibodies), immunotherapy (e.g.anti-PD-1 antibody,anti-PD-L1 antibody,anti-PD-L2 antibody or CTLA-4 antibody),or other clinical trials agents;
9. No limit to previous endocrine therapy.
10. Age between 18 and 75 years;
11. ECOG performance status of 0 or 1;
12. Life expectancy: more than 2 years;
13. Hematopoietic: WBC>3×109/L;PLT>80×109/L; Hb>90g/L;
14. Hepatic: ALT and AST<2 times upper limit of normal (ULN); bilirubin<1.5 times ULN;
15. Renal: creatinine <1.5 times ULN or creatinine clearance ≥ 60 mL/min.

Exclusion Criteria:

1. Arrhythmias require antiarrhythmic therapy (with the exception of β-blockers or digoxin), symptomatic coronary artery disease or local myocardial ischemia (myocardial infarction within the past 6 months) or congestive heart failure exceeding NYHA II;
2. Severe hypertension with poor control after medication;
3. A known history of testing positive for HIV or chronic hepatitis B or C (high copy virus DNA) at active stage;
4. Patients with active tuberculosis (TB) are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year before screening;
5. Other active severe clinical infections (NCI-CTC5.0);
6. Apparent distant metastasis away from the pelvic before surgery;
7. Cachexia, organ function decompensation;
8. Previous pelvic or abdominal radiotherapy;
9. Multiple primary colorectal cancers;
10. Epilepsy require medical treatment (such as steroid or antiepileptic therapy);
11. Other malignancy within the past 5 years with the exception of effectively treated carcinoma in situ of the cervix or basal cell carcinoma of the skin;
12. Drug abuse and medical, psychological or social factors that may interfere with patients' participation in the study or affect the evaluation of the study;
13. Patients have any active autoimmune diseases or a history of autoimmune diseases(including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism and decreased thyroid function; patients with vitiligo or with complete remission of asthma in childhood and without any intervention in adulthood may be included; patients with asthma requiring bronchodilators intervention are not included.
14. Received any anti-infection vaccine (e.g. influenza vaccine, chickenpox vaccine, etc.) within 4 weeks before enrollment;
15. Complications require long-term treatment with immunosuppressive drugs, or requiring systemic or local use of immunosuppressive corticosteroids(>10mg/day prednisone or other therapeutic hormones);
16. Known or suspected allergy to the study drugs or to any drugs related to this trial;
17. Any unstable condition or which endangers the patients' safety and compliance;
18. Pregnant or breast-feeding women who are fertile without effective contraception;
19. Refuse to sign the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2026-10-18 (Estimated); Study Completion 2026-10-18 (Estimated)

PRIMARY OUTCOMES:
complete response rate | 6 weeks after curative surgery for pCR; 6 weeks after the completion of neoadjuvant therapy for cCR
  the proportion of CR cases (pCR for those who underwent surgery and cCR for those who didn't receive surgery)

SECONDARY OUTCOMES:
Acute toxiticy according CTCAE5.0 | From start of treatment to 3 months after the adjuvant therapy or last dose of treatment
  Acute toxiticy according CTCAE5.0
Tumor regresssion grade according to AJCC TRG grading system | 6 weeks after curative surgery
  Tumor regresssion grade according to AJCC TRG grading system
R0 resection rate | 6 weeks after curative surgery
  R0 resection rate
Local recurrence | 5 years after curative surgery
  Local recurrence
Distant metastasis | 5 years after curative surgery
  Distant metastasis
Tumor response | 6 weeks after first study treatment
  tumor volume reduction rate (TVRR) reaching 20% or above

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Oncology,Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Allegra CJ, Yothers G, O'Connell MJ, Beart RW, Wozniak TF, Pitot HC, Shields AF, Landry JC, Ryan DP, Arora A, Evans LS, Bahary N, Soori G, Eakle JF, Robertson JM, Moore DF Jr, Mullane MR, Marchello BT, Ward PJ, Sharif S, Roh MS, Wolmark N. Neoadjuvant 5-FU or Capecitabine Plus Radiation With or Without Oxaliplatin in Rectal Cancer Patients: A Phase III Randomized Clinical Trial. J Natl Cancer Inst. 2015 Sep 14;107(11):djv248. doi: 10.1093/jnci/djv248. Print 2015 Nov. PMID 26374429
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Derived] Chen G, Jin Y, Guan WL, Zhang RX, Xiao WW, Cai PQ, Liu M, Lin JZ, Wang FL, Li C, Quan TT, Xi SY, Zhang HZ, Pan ZZ, Wang F, Xu RH. Neoadjuvant PD-1 blockade with sintilimab in mismatch-repair deficient, locally advanced rectal cancer: an open-label, single-centre phase 2 study. Lancet Gastroenterol Hepatol. 2023 May;8(5):422-431. doi: 10.1016/S2468-1253(22)00439-3. Epub 2023 Mar 1. PMID 36870360